CLINICAL TRIAL: NCT03923868
Title: A Randomized, Double-blind, Placebo-controlled, Multiple-administration, Multiple-dose, Phase Ib/IIa Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of D-0120 Tablets in Healthy Subjects and Hyperuricemia Patients in China
Brief Title: D-0120 Safety and PK/PD Study in China
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: IBIO-202
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Hyperuricemia or Gout
MeSH Terms: conditions — Hyperuricemia; Gout

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- dose escalation in healthy subjects (Experimental)
  Interventions: Drug: D-0120
- dose escalation in hyperuricemia patients (Experimental)
  Interventions: Drug: D-0120

INTERVENTIONS:
Drug: D-0120 — D-0120 monotherapy dose escalation, oral, multiple dose for up to 28 days

SUMMARY:
It is a randomized, double-blind, placebo-controlled, multiple-administration, multiple-dose, dose-escalating, phase Ib/IIa clinical study to evaluate the safety, tolerability, PK and PD of D-0120 in healthy subjects and hyperuricemia patients (gout or asymptomatic) in China.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old and ≤ 65 years old;
2. Phase Ib: fasting sUA in the morning of screening period (fasted after 8:00 pm on the previous day) of healthy subjects meets the following requirement: 270 umol/l (4.5 mg/dL) ≤ sUA <420 umol/l (7 mg/dL)

   Phase IIa: hyperuricemia subjects should meet any of the following:
3. Subject's BMI range is 18.0~32.0 kg/m2 (inclusive);
4. Female subjects must be non-pregnant and non-lactating, surgically sterilized or ≥ 60 years old. Male subjects must be surgically sterilized or agree to practice sexual abstinence;
5. Results of routine blood tests, blood biochemical tests and routine urine tests are within the normal range or clinically insignificant as judged by the principle investigator. Routine urine tests include normal urine creatinine, urine protein/creatinine ratio. ECGs are within the normal range or clinically insignificant as judged by the principle investigator.
6. Subjects have the ability to follow study and follow-up procedures.
7. Subjects have the ability to understand the study protocol and the risks involved, and must provide signed informed consent form to participate in the study.

Exclusion Criteria:

1. History of significant metabolic, hematological, pulmonary, cardiovascular, gastrointestinal, nervous, hepatic, renal, urinary, gastrointestinal, immune, endocrine, psychiatric diseases, or clinical abnormalities that may pose excessive risks to the subjects or affect outcome or study interpretation at the discretion of the investigators;
2. Allergic constitution, or allergy to any drug used in the study or any ingredient of study drug;
3. History of malignant tumors;
4. Subjects with positive results of any of the following items: screening hepatitis C antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab), hepatitis B surface antigen (HBsAg) and treponema pallidum (only for phase Ib healthy subjects);
5. Urinary calculi confirmed by B-ultrasound during screening period;
6. Myocardial infarction, angina pectoris, percutaneous transluminal coronary angioplasty, coronary artery bypass grafting, cerebral infarction, cerebral hemorrhage, subarachnoid hemorrhage or transient ischemic attack within 3 months prior to screening;
7. Participation in clinical studies of any investigational drugs or medical devices within 3 months prior to screening;
8. Major surgery within 3 months prior to randomization;
9. Any clinically significant acute diseases within one month prior to screening at the discretion of the investigators;
10. Gout flare within 14 days prior to randomization;
11. Use of other uric acid-lowering drugs (allopurinol, febuxostat, probenecid, benzbromarone) within 14 days prior to randomization;
12. Daily dose of aspirin > 100 mg within 14 days before randomization;
13. Use of any diuretic within 14 days before randomization;
14. Use of any Chinese herbal medicine within 14 days before randomization;
15. History of drug abuse or alcohol abuse (for phase Ib healthy subjects, the screening alcohol test and urine drug test are positive);
16. Any situation that may prevent the subject from completing the study or pose a significant risk to the subject as considered by any investigator;
17. Any other situation that may pose excessive risks to the subject or affect outcome or study interpretation as considered by any investigator;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The number of subjects with treatment-related adverse events as assessed | Day 1 - Day 28
  Data will include clinical observations, ECG parameters, clinical chemistry and haematology and vital signs assessed as the number of subjects with treatment-related adverse events assessed

SECONDARY OUTCOMES:
Time to observed Cmax (Tmax) for D-0120 | Day 1 - Day 28
  Blood samples will be collected to assess plasma concentrations of D-0120 at a series of timepoints to derive Tmax
Area under the plasma concentration-time curve (AUC) for D-0120 | Day 1 - Day 28
  Blood samples will be collected to assess plasma concentrations of D-0120 at a series of timepoints to derive AUC
Maximum Observed Plasma Concentration (Cmax) of D-0120 | Day 1 - Day 28
  Blood samples will be collected to assess plasma concentrations of D-0120 at a series of timepoints to derive Cmax

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Site 04, Bengbu, Anhui
  - Site 03, Nanjing, Jiangsu
  - Site 07, Nanjing, Jiangsu
  - Site 01- The second affiliated hospital of zhejiang university school of medicine, Hangzhou, Zhejiang
  - Site 06, Huzhou, Zhejiang
  - Site 05, Wenzhou, Zhejiang